CLINICAL TRIAL: NCT04026425
Title: Probing Metabolism, Circulating Inflammatory Molecules, Extracellular Vesicles and Immune Dysregulation in Individual Immune Cells in ME/CFS
Brief Title: Analysis of Post-exertional Malaise Using a Two-day CPET in People With ME/CFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ithaca College (Other)
Collaborators: Cornell University (Other); Weill Medical College of Cornell University (Other); Workwell Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: U54NS105541 (NIH); 5U54NS105541 (NIH)
Record Dates: First submitted 2019-07-02; First posted 2019-07-19 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome
Keywords: cardiopulmonary exercise test (CPET); post-exertional malaise (PEM)
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ME/CFS (Experimental): Adults with ME/CFS
  Interventions: Other: Two-day cardiopulmonary exercise test
- Healthy controls (Active Comparator): Healthy, low-active adults
  Interventions: Other: Two-day cardiopulmonary exercise test

INTERVENTIONS:
Other: Two-day cardiopulmonary exercise test — A series of two cardiopulmonary exercise tests (CPETs) performed over two days. Participants will perform a CPET and then will return approximately 24 hours later to perform the second CPET. The CPET begins with 3 minutes of seated rest followed by cycling during incremental workloads which increases 15 watts throughout each minute of exercise. The participant will cycle until volitional exhaustion and/or the participant and/or test administrator determines to stop the test. Actual exercise time usually varies between 8-10 minutes.

SUMMARY:
This study aims to collect and identify key outcome measures or disease parameters in ME/CFS that are altered during elevated symptoms relative to baseline by gathering information before and after symptom provocation using a two-day cardiopulmonary exercise test.

DETAILED DESCRIPTION:
The phenomenon of post-exertional malaise (PEM), in which an ME/CFS patient's symptoms are elevated following even low-level exertion, is a hallmark feature of the disease. The cause of PEM, like the cause of ME/CFS, is not understood. This study aims to utilize a two-day CPET to invoke PEM. This provides a unique opportunity to collect data on how key outcome measures or disease parameters are altered during elevated symptoms relative to baseline within each patient by gathering information before and after symptom provocation.

A total of 90 participants and 90 controls will undergo CPET testing. Participation will be split amongst three different sites (Ithaca, NY, New York, NY, and Los Angeles, CA). Subjects will be located in urban and rural areas to establish relatively diverse study populations.

This study is a component of the Cornell ME/CFS Collaborative Research Center (CRC). Blood samples taken before and after CPET will be utilized in associated projects with the Cornell ME/CFS CRC. CPET data along with the analysis of blood samples has great potential to reveal why exercise negatively affects ME/CFS patients and thus perhaps why patients are also impaired even before increasing their activity level.

ELIGIBILITY:
Adults with ME/CFS:

Inclusion Criteria:

* Diagnosed with ME/CFS
* Adults 18 to 70 years of age

Exclusion Criteria:

* Recent history of panic attacks within the past 6 months
* Diagnosis of schizophrenia, major depressive disorder, bipolar disorder, or an anxiety disorder such as OCD or PTSD
* Hospitalized for a psychological condition within the last 6 months
* Unwilling to stop taking nutritional supplements, including probiotics, two weeks before the exercise tests.
* Unwilling to stop pain medication and stimulant medication two days before the exercise tests.
* Smoker, or stopped smoking less than 1 year ago
* Pregnant or breastfeeding
* Diabetic
* Have an orthopedic limitation that prohibits cycle exercise
* Excessive alcohol consumption

Healthy Volunteers:

Inclusion Criteria:

* Healthy
* Low-active
* Adults 18 to 70 years of age

Exclusion Criteria:

* Recent history of panic attacks within the past 6 months
* Diagnosis of schizophrenia, major depressive disorder, bipolar disorder, or an anxiety disorder such as OCD or PTSD
* Hospitalized for a psychological condition within the last 6 months
* Unwilling to stop taking nutritional supplements, including probiotics, two weeks before the exercise tests.
* Unwilling to stop pain medication and stimulant medication two days before the exercise tests.
* Smoker, or stopped smoking less than 1 year ago
* Pregnant or breastfeeding
* Diabetic
* Have an orthopedic limitation that prohibits cycle exercise
* Excessive alcohol consumption

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Volume of oxygen consumed at peak effort | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  Volume of oxygen consumed at peak effort during CPET 1 and during CPET 2.
Volume of oxygen consumed at ventilatory/anaerobic threshold (VAT) | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  VAT is a non-invasive surrogate measure for anaerobic threshold, which is indicated during incremental exercise by a non-linear increase in rate of carbon dioxide production relative to rate of oxygen consumption.
Rate of work performed at peak effort | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  Rate of work performed at peak effort during CPET 1 and during CPET 2. Rate of work is measured in Watts.
Rate of work performed at VAT | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  Rate of work performed at VAT during CPET 1 and during CPET 2. Rate of work is measured in Watts.
Heart rate at peak effort | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  Heart rate at peak effort during CPET 1 and during CPET 2.
Heart rate at VAT | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  Heart rate at VAT during CPET 1 and during CPET 2.
Systolic blood pressure at seated rest | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  Systolic blood pressure at seated rest 1-minute before the start of CPET 1 and 1-minute before the start of CPET 2.
Systolic blood pressure at peak effort | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  Systolic blood pressure at peak effort during CPET 1 and during CPET 2.
Respiratory Exchange Ratio (RER) at peak effort | During intervention on day 1 and during intervention on day 2; assessed through study completion, approximately 4 years from study start date.
  RER at peak effort during CPET 1 and during CPET 2. RER is calculated as the rate of carbon dioxide production divided by the rate of oxygen consumption, and during exercise is an indicator of participant effort.

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Keller, Ph.D., Study Director — Ithaca College; Geoff Moore, M.D., Study Director — Ithaca College
Locations (3):
- United States (3):
  - ID Med, Torrance, California
  - Ithaca College, Ithaca, New York
  - Weill Cornell Medicine, New York, New York

REFERENCES:
- [Derived] Keller B, Receno CN, Franconi CJ, Harenberg S, Stevens J, Mao X, Stevens SR, Moore G, Levine S, Chia J, Shungu D, Hanson MR. Cardiopulmonary and metabolic responses during a 2-day CPET in myalgic encephalomyelitis/chronic fatigue syndrome: translating reduced oxygen consumption to impairment status to treatment considerations. J Transl Med. 2024 Jul 5;22(1):627. doi: 10.1186/s12967-024-05410-5. PMID 38965566
- See also: Related information — https://neuroimmune.cornell.edu/research/